CLINICAL TRIAL: NCT06287346
Title: 5-Years Multicentric Prospective Post-Market Clinical Follow-up (PMCF) Comparative Study of CeraRoot Ceramic Dental Implants One-piece Versus Two-piece.
Brief Title: 5-Years PMCF Study of Ceramic Dental Implants One-piece Versus Two-piece.
Acronym: 240101
Status: Recruiting | Type: Observational
Sponsor: CeraRoot SL (Industry)
Responsible Party: Sponsor
Other Study IDs: 240101
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Edentulism; Tooth Loss
Keywords: dental implant; ceramic dental implant; zirconia implant; y-tzp; metal-free
MeSH Terms: conditions — Tooth Loss | interventions — Dental Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- One-piece: One-piece CeraRoot dental implants
  Interventions: Device: dental implant
- Two-piece (TL): Two-piece CeraRoot TL dental implants
  Interventions: Device: dental implant

INTERVENTIONS:
Device: dental implant — ceramic dental implant

SUMMARY:
The goal of this cohort observational study is to compare in the survival rate of ceramic dental implants placed in patients with missing or hopeless teeth . The main question[s] it aims to answer are:

* Are there any significant differences in survival rate between the use of one-piece ceramic implant versus the two-piece (TL) variant?
* What are the complications associated to the procedure and differences between the two groups.

DETAILED DESCRIPTION:
The present clinical study protocol has the objective to compare the performance of different CeraRoot ceramic implant models (16,11,21,12,14,34,34L) and the different sub-variants (one-piece versus two-piece).

The geographic population of study will be the patients in two different dental centers located in Barcelona (Spain) and Boulder (Colorado, USA). The intended population as described in the device instruction for use (3) is " Intended Population: All fully-grown patients (men or women) requiring dental reconstruction using dental implants and who have no contraindications. The CeraRoot® dental implants are specially indicated in patients with metal allergies and chronic illness due to metal allergies.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of partial or total edentulism.
* Specially indicated for patients with metal allergies and chronic illness due to metal allergies.

Exclusion Criteria:

1. General Contraindications:

   1. Local and Systemic contraindications for surgery.
   2. Poor oral hygiene
   3. Patients with health problems, disease or any physical or psychological condition to which an oral surgery may be contraindicated.
2. Relative Contraindications:

   1. Previously irradiated bone
   2. diabetes
   3. anticoagulant medication
   4. hemodynamic problems
   5. bruxism
   6. Para functional habits
   7. bad bone anatomy
   8. smokers
   9. none controlled periodontitis
   10. malocclusions
   11. TMJ problems
   12. diseases in the oral cavity
   13. pregnancy
   14. insufficient oral hygiene for adequate health.
3. Local contraindications

   1. insufficient bone quantity or quality
   2. remaining of roots
   3. localized periodontal disease
   4. Any pathology in the neighboring teeth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The geographic population of study will be the patients in two different private dental centers located in Barcelona (Spain) and Boulder (Colorado, USA).
Sampling Method: Non-Probability Sample
Enrollment: 652 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Survival rate | From enrolment to the end of treatment 12 months or more.
  The implant is osseointegrated and in function in the patient's jaw without pain and no mobility.

SECONDARY OUTCOMES:
Complications | 1 year after treatment
  Implantitis, mucositis, pain, implant fracture, prosthetic fracture, bone loss,

CONTACTS AND LOCATIONS:
Locations (2):
- Family Holistic Dentistry, Boulder, Colorado, United States
- CeraRoot CLINIC, Les Franqueses del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
at the end of the study the results will be published including, method and results survival rates and complications rate. For this reason no need to share any other information

REFERENCES:
- [Background] undefined